CLINICAL TRIAL: NCT03077555
Title: Ovulation and Follicular Development Associated With Mid Follicular Phase Initiation of Combined Hormonal Contraception Containing Estradiol Hemihydrate Compared to Ethinyl Estradiol
Brief Title: Ovulation and Follicular Development Associated With Mid Follicular Phase Initiation of Combined Hormonal Contraception
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Preeyaporn Jirakittidul, Principle investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Si804/2016
Record Dates: First submitted 2017-03-02; First posted 2017-03-13 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Ovulation Inhibition
Keywords: quick starting contraception

STUDY DESIGN:
Intervention Model Description: two intervention groups
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meliane ED (Active Comparator): 20 mcg ethinyl estradiol/70 mcg gestodene
  Interventions: Drug: Meliane ED
- Zoely (Experimental): 1.5 mg estradiol/2.5 mg nomegestrol acetate
  Interventions: Drug: Zoely

INTERVENTIONS:
Drug: Zoely — quick start of combined hormonal contraception containing 1.5 mg estradiol /2.5 mg nomegestrol acetate
  Other Names: estradiol hemihydrate combined pills
  Arms: Zoely
Drug: Meliane ED — quick start of combined hormonal contraception containing 20 mcg ethinyl estradiol /75 mcg gestodene
  Other Names: ethinyl estradiol combined pills
  Arms: Meliane ED

SUMMARY:
Quick starting combined oral contraception containing estradiol hemihydrate/nomegestrol acetate is effective to inhibit ovulation in healthy reproductive age women and non-inferiority to combined oral contraception containing ethinyl estradiol/gestodene.

DETAILED DESCRIPTION:
This study is a randomized control, non-inferiority trial which compare the proportion of ovulation between two oral combined pills when delay starting the first tablet at mid-follicular phase of menstrual cycle in 18 - 40 year old, healthy women with prior normal and regular periods. Participations will be undergone trans-vaginal or trans-rectal ultrasonography between day 1 - 3 of menstrual period for evaluation of ovarian follicle/cyst (if present). Only women who have normal looking of ovaries without dominant ovarian follicle will be included in study-protocol. Immediately after trans-vaginal/trans-rectal ultrasound between day 7 - 9 of menstrual period, all participants will be randomly assigned to receive one pack of investigated pills (1.5 mg estradiol hemihydrate/2.5 mg nomegestrol acetate or 20 mcg ethinyl estradiol/75 mcg gestodene) and to take the first tablet under direct observation by research-nurse. Participants will take one consecutive tablet at about the same time each day until complete pack. The next appointments will be every 2 - 3 days to monitor ovarian function by using Hoogland score until ovulation or follicular quiescence will be presented. The last visit will be about 1 week after complete pack to monitor adverse effect and safety through out the protocol.

ELIGIBILITY:
Inclusion Criteria:

* healthy women, age 18 - 40 years
* prior normal and regular interval of menstruation

Exclusion Criteria:

* current breast feeding women
* within 1 month period of child-delivery or miscarriage
* body mass index 30 kg/m2 or more
* contraindicated to use combined hormonal contraception
* current using other hormonal drugs that affect ovulation function

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 69 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
ovulation inhibition | 1 month
  comparison of ovulation inhibition effect between Zoely and Meliane ED with mid follicular phase starting

SECONDARY OUTCOMES:
follicular development | through study completion, an average of 1 month
  pattern of ovarian follicular change after receive intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Undecided